CLINICAL TRIAL: NCT05581745
Title: Blood Group A2 Donor to Blood Group O Recipient Lung Transplantation
Brief Title: A2 to O Lung Transplants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-5005
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Lung Transplant; ABO Incompatibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A2 donor transplant to O recipient (Experimental)
  Interventions: Procedure: Blood group A2 donor to blood group O recipient lung transplant surgery

INTERVENTIONS:
Procedure: Blood group A2 donor to blood group O recipient lung transplant surgery — Suitable blood group A2 donor lung transplant to a consented blood group O recipient who has acceptably low levels of anti-A antibody titres and a negative virtual cross-match at time of transplant

SUMMARY:
Blood group A2 to blood group O kidney and liver transplants have been shown to be safe and successful, especially in recipients with low pre-operative anti-A antibody titers and with the use of peri-operative antibody-depleting therapies. Since blood group O lung transplant candidates tend to have longer wait times and a higher waitlist mortality compared to other blood groups, we propose to conduct a prospective study of lung transplantation from blood group A2 donors to eligible blood group O recipients in an effort to increase the available donor pool. The aim of this study is to determine both the feasibility and safety of this specific type of ABO-incompatible lung transplant, and the impact of this practice on reducing transplant wait times among blood group O lung transplant candidates. This would represent the first prospective study of ABO-incompatible lung transplants worldwide.

ELIGIBILITY:
Inclusion Criteria:

* first lung transplant
* blood group O recipient
* low pre-operative anti-A antibody titers
* consent to study participation

Exclusion Criteria:

* re-transplant
* multiorgan transplant
* positive virtual crossmatch at time of transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-transplant anti-A antibody titers | post-op day 5 or day 12
Primary graft dysfunction grade | post-op day 0, 1, 2, 3
Incidence of hyperacute antibody-mediated rejection | post-op day 1, 2
C4d positivity on transbronchial biopsy samples | 1 year
Incidence and severity of acute cellular rejection | 1 year
Bleeding | post-op day 1-7
Infection | 10 years
Graft function | 10 years
Incidence of malignancy | 10 years
Chronic lung allograft dysfunction | 10 years
Time to death or re-transplantation | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Shaf Keshavjee, MD MSc FRCSC FACS, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada